CLINICAL TRIAL: NCT00520299
Title: Phase 1/2 Study of ADI-SS PEG 20,000mw in Patients With Advanced Melanoma
Brief Title: Study of ADI-PEG 20 in Patients With Advanced Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2005-007; MSKCC IRB #06-165 (Other: MSKCC IRB); NYU IRB #07-053 (Other: NYU School of Medicine IRB)
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Melanoma; Skin Cancer; Neoplasm
Keywords: metastatic melanoma; ADI; ADI-PEG 20; ADI SS PEG 20,000mw; arginine; enzyme therapy
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Neoplasms | interventions — ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Subjects received ADI-PEG 20 at a dose of 40 IU/m^2
  Interventions: Drug: ADI PEG 20
- Cohort 2 (Experimental): Subjects received ADI-PEG 20 at a dose of 80 IU/m^2
  Interventions: Drug: ADI PEG 20
- Cohort 3 (Experimental): Subjects received ADI-PEG 20 at a dose of 160 IU/m^2
  Interventions: Drug: ADI PEG 20

INTERVENTIONS:
Drug: ADI PEG 20 — Intramuscular injections were administered into the deltoid, gluteal, or quadricep muscles once weekly (± 2 days) for 9 weeks during cycle 1 and 8 weeks during subsequent cycles
  Other Names: ADI-SS PEG 20,000 mw; ADI

SUMMARY:
This was a phase 1/2, open-label, dose-escalation study of arginine deiminase linked via succinimidyl succinate to polyethylene glycol of 20,000 molecular weight (ADI-PEG 20) in subjects with advanced melanoma. ADI-PEG 20 was administered intramuscularly (IM) at escalating doses weekly for 9 weeks (cycle 1) or 8 weeks (subsequent cycles). The primary objectives were to the establish the safety, tolerability, and clinical efficacy of ADI-PEG 20. Secondary objectives included evaluation of the metabolic activity by [18F]-fluorodeoxyglucose positron emission tomography (FDG PET), pharmacodynamics, correlation of immunogenicity with clinical response, and correlation of argininosuccinate synthetase (ASS) tumor expression with clinical response.

DETAILED DESCRIPTION:
A 3+3 design was implemented during phase 1, in which 3 to 6 subjects were enrolled sequentially into the following escalating dose cohorts:

* Cohort 1 (40 IU/m^2)
* Cohort 2 (80 IU/m^2)
* Cohort 3 (160 IU/m^2)

Subjects were monitored for dose-limiting toxicity (DLT) during the first 2 weeks of cycle 1, with DLT defined as any grade 3 or higher toxicity. The maximum tolerated dose (MTD) was defined as the cohort in which < 33% of subjects (ie, 0/3 or 1/6 subjects in a cohort) experienced DLT. In phase 2, the MTD cohort was expanded in up to 25 patients.

Subjects who completed treatment in cycle 1 without DLT were eligible to initiate cycle 2 at week 10 provided that a computed tomography (CT) scan showed either enlargement of existing disease without accompanying symptoms OR stable disease or improvement with no unacceptable toxicity. The same radiologic criteria applied for initiation of subsequent cycles. Subjects could continue to receive study treatment until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed malignant melanoma, American Joint Committee on Cancer (AJCC) stage III (unresectable) or IV. Subjects with uveal and mucosal melanomas were eligible.
2. Measurable disease using the Response Evaluation Criteria in Solid Tumors (RECIST).
3. Pathology slides reviewed by the Memorial Hospital Department of Pathology or New York University (NYU) Department of Pathology for confirmation of melanoma diagnosis.
4. Karnofsky performance status of 80% or more.
5. Adequate organ and marrow function, as defined below:

   * white blood cell count ≥ 3000/µL
   * absolute neutrophil count ≥ 1500/µL
   * platelet count ≥ 100,000/µL
   * total bilirubin ≤ 2.5 x institutional upper limit of normal (ULN)
   * lactate dehydrogenase ≤ 1.5 x institutional ULN
   * albumin ≥ 3.0 mg/dL
   * creatinine ≤ 2.0 mg/dL
6. Expected survival of at least 3 months.
7. Age ≥ 18 years.
8. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Receipt of chemotherapy, immunotherapy, or radiotherapy within 3 weeks prior to first dosing of study agent or lack of recovery from adverse events (AEs) due to agents administered more than 3 weeks earlier. For nitrosoureas, at least 6 weeks must have elapsed.
2. Any other malignancy that required concomitant therapy.
3. Any medical condition that could have made it difficult for the subject to complete the full course of treatments, at the discretion of the Principal Investigator or co-Principal Investigators.
4. Metastatic disease to the central nervous system, unless treated and stable.
5. Known human immunodeficiency virus (HIV) positivity.
6. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
7. Lack of availability for clinical follow-up assessments.
8. Participation in any other clinical trial involving another investigational agent within 3 weeks prior to enrollment.
9. Pregnant women or women who were nursing. Women of child-bearing potential and sexually active men must have used appropriate contraception during the course of this study. Women of child-bearing potential must not have been pregnant (negative β human chorionic gonadotropin within 2 weeks of treatment) or nursing during treatment.
10. History of seizure disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jedd Wolchok, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Anna Pavlick, DO, Principal Investigator — New York University Cancer Institute; Gary Schwartz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - NYU Cancer Institute, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ott PA, Carvajal RD, Pandit-Taskar N, Jungbluth AA, Hoffman EW, Wu BW, Bomalaski JS, Venhaus R, Pan L, Old LJ, Pavlick AC, Wolchok JD. Phase I/II study of pegylated arginine deiminase (ADI-PEG 20) in patients with advanced melanoma. Invest New Drugs. 2013 Apr;31(2):425-34. doi: 10.1007/s10637-012-9862-2. Epub 2012 Aug 5. PMID 22864522

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: ADI-PEG 20 40 IU/m^2/Week: Includes subjects enrolled to receive 40 IU/m^2/week of ADI-PEG 20
- Cohort 2: ADI-PEG 20 80 IU/m^2/Week: Includes subjects enrolled to receive 80 IU/m^2/week of ADI-PEG 20
- Cohort 3: ADI-PEG 20 160 IU/m^2/Week: Includes subjects enrolled to receive 160 IU/m^2/week of ADI-PEG 20
Period: Overall Study
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Started | 6 | 6 | 19
Completed | 6 (Defined as completion of 1 treatment cycle) | 3 | 13
Not Completed | 0 | 3 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Progressive disease | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (all subjects who received at least 1 dose of ADI-PEG 20)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week | Total
Number analyzed (Participants) | 6 | 6 | 19 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (18.2) | 61.2 (14.7) | 67.2 (11.2) | 64.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 6 | 14
  Male | 1 | 3 | 13 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 17 | 29
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 6 | 18 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.0 (4.1) | 24.7 (1.8) | 26.9 (4.7) | 25.5 (4.5)
ASS Assay Result [Number; unit: participants] — Argininosuccinate synthetase (ASS) tumor expression, as determined by immunohistochemistry, is categorized as either negative or ≤ 5% positive tumor cells.
  participants
    Negative | 4 | 6 | 14 | 24
    ≤5% positive | 2 | 0 | 3 | 5
    Not done | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Safety and Tolerability of ADI-PEG 20
Description: Analysis of treatment-emergent adverse events (TEAEs) reported from clinical laboratory tests, physical examinations, and vital signs.
Time Frame: Every 1 to 2 weeks for up to 12 months
Population: Safety Analysis Set (all subjects who received at least 1 dose of ADI-PEG 20)
Measure: Number; unit: participants
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Number analyzed (Participants) | 6 | 6 | 19
participants
  Any TEAE | 6 | 6 | 19
  Grade 3 TEAE | 1 | 2 | 4
  Grade 4 TEAE | 0 | 1 | 1
  Grade 5 TEAE (Death) | 0 | 0 | 1
  Treatment-related TEAE | 5 | 5 | 17
  SAE | 4 | 1 | 6
  TEAE leading to withdrawal | 0 | 1 | 3

2. Primary Outcome: Best Overall Clinical Tumor Response
Description: Clinical tumor responses were evaluated using disease imaging (CT preferred) performed at baseline and at the end of every cycle. Responses were categorized according to RECIST. Per RECIST for target lesions and assessed by MRI: Complete Response (CR): Disappearance of all target lesions [no evidence of disease]; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Every 8 to 9 weeks for up to 12 months
Population: Includes all subjects who completed the study as planned or had tumor progression during the study
Measure: Number; unit: participants
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Number analyzed (Participants) | 6 | 6 | 17
participants
  Complete/partial response | 0 | 0 | 0
  Stable disease | 3 | 2 | 4
  Progressive disease | 3 | 4 | 13

3. Secondary Outcome: Metabolic Tumor Response
Description: Metabolic tumor responses were evaluated using fluorodeoxyglucose (FDG) positron emission tomography (PET) at baseline, on day 4, and at the end of every cycle.
Time Frame: Every 8 to 9 weeks for up to 12 months
Population: Includes all subjects who completed the study as planned or had tumor progression during the study
Measure: Number; unit: participants
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Number analyzed (Participants) | 6 | 6 | 17
participants
  Cycle 1 Day 4: Partial metabolic response | 1 | 0 | 6
  Cycle 1 Day 4: Stable metabolic disease | 2 | 3 | 6
  Cycle 1 Day 4: Progressive metabolic disease | 3 | 2 | 4
  Cycle 1 Day 4: Missing | 0 | 1 | 1
  Cycle 1 Day 50: Partial metabolic response | 0 | 1 | 0
  Cycle 1 Day 50: Stable metabolic disease | 4 | 3 | 5
  Cycle 1 Day 50: Progressive metabolic disease | 2 | 1 | 9
  Cycle 1 Day 50: Missing | 0 | 1 | 3

4. Secondary Outcome: Summary of ADI-PEG 20 Plasma Concentrations Over Time
Description: Blood samples were collected on day 1 (pre-injection), day 4, day 8, and every 7 days thereafter for ADI-PEG 20 plasma concentrations.
Time Frame: Up to 12 months
Population: Includes all subjects who had at least 1 post-baseline blood sample with associated pharmacokinetic analysis. Means are presented for time points at which >1 subject in any arm contributed data.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Number analyzed (Participants) | 6 | 5 | 19
nM
  Day 0: number analyzed (Participants) | 6 | 5 | 10
  Day 0 | 3.3 (2.9) | 4.4 (5.2) | 1.9 (1.7)
  Day 4 | 35.5 (16.0) | 59.8 (35.7) | 57.2 (39.9)
  Day 8 | 33.2 (17.2) | 46.3 (33.8) | 60.9 (35.5)
  Day 15: number analyzed (Participants) | 6 | 5 | 18
  Day 15 | 37.7 (27.2) | 49.8 (59.4) | 54.0 (36.4)
  Day 22: number analyzed (Participants) | 6 | 5 | 18
  Day 22 | 24.1 (16.9) | 61.2 (63.8) | 47.5 (40.2)
  Day 29: number analyzed (Participants) | 5 | 5 | 16
  Day 29 | 16.8 (11.1) | 54.0 (58.2) | 40.9 (42.3)
  Day 36: number analyzed (Participants) | 6 | 5 | 15
  Day 36 | 11.2 (11.7) | 50.0 (65.3) | 27.1 (42.3)
  Day 43: number analyzed (Participants) | 6 | 5 | 14
  Day 43 | 12.0 (10.7) | 34.9 (47.2) | 11.9 (20.2)
  Day 50: number analyzed (Participants) | 6 | 5 | 14
  Day 50 | 11.0 (14.9) | 19.0 (26.2) | 13.2 (25.7)
  Day 57: number analyzed (Participants) | 6 | 5 | 14
  Day 57 | 8.4 (10.5) | 9.3 (10.3) | 10.0 (15.6)
  Day 64: number analyzed (Participants) | 5 | 3 | 11
  Day 64 | 8.0 (9.1) | 14.7 (17.3) | 10.0 (16.2)
  Day 71: number analyzed (Participants) | 3 | 2 | 4
  Day 71 | 2.6 (1.3) | 1.5 (0.7) | 3.8 (2.9)
  Day 78: number analyzed (Participants) | 3 | 2 | 4
  Day 78 | 2.8 (1.1) | 0.6 (0.8) | 2.6 (1.2)
  Day 85: number analyzed (Participants) | 3 | 2 | 4
  Day 85 | 0.5 (0.7) | 0.2 (0.0) | 2.2 (1.9)
  Day 92: number analyzed (Participants) | 3 | 2 | 4
  Day 92 | 0.9 (0.8) | 0.6 (0.4) | 2.6 (2.9)
  Day 99: number analyzed (Participants) | 3 | 1 | 4
  Day 99 | 0.9 (1.1) | 2.2 (NA) — Only 1 participant contributed data at this time point. | 2.4 (1.7)
  Day 106: number analyzed (Participants) | 3 | 1 | 4
  Day 106 | 1.0 (1.7) | 3.1 (NA) — Only 1 participant contributed data at this time point. | 0.9 (0.8)
  Day 113: number analyzed (Participants) | 2 | 1 | 4
  Day 113 | 0.9 (0.1) | 2.0 (NA) — Only 1 participant contributed data at this time point. | 1.6 (1.8)
  Day 120: number analyzed (Participants) | 2 | 1 | 4
  Day 120 | 2.1 (0.7) | 3.0 (NA) — Only 1 participant contributed data at this time point. | 4.0 (2.4)

5. Secondary Outcome: Summary of Plasma Arginine Levels Over Time
Description: Blood samples were collected at baseline, day 1 (pre-injection), day 4, day 8, and every 7 days thereafter for plasma arginine levels.
Time Frame: Up to 9 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Number analyzed (Participants) | 6 | 5 | 19
uM
  Day 0: number analyzed (Participants) | 6 | 5 | 10
  Day 0 | 55 (17) | 62 (22) | 49 (11)
  Day 4 | 2 (0) | 9 (20) | 4 (11)
  Day 8 | 2 (0) | 12 (18) | 3 (7)
  Day 15: number analyzed (Participants) | 6 | 5 | 18
  Day 15 | 4 (6) | 29 (22) | 7 (16)
  Day 22: number analyzed (Participants) | 6 | 5 | 18
  Day 22 | 9 (11) | 22 (23) | 21 (33)
  Day 29: number analyzed (Participants) | 5 | 5 | 16
  Day 29 | 14 (24) | 19 (24) | 23 (32)
  Day 36: number analyzed (Participants) | 6 | 5 | 15
  Day 36 | 20 (28) | 29 (26) | 31 (34)
  Day 43: number analyzed (Participants) | 6 | 5 | 14
  Day 43 | 23 (34) | 35 (31) | 48 (44)
  Day 50: number analyzed (Participants) | 6 | 5 | 14
  Day 50 | 58 (46) | 24 (21) | 44 (37)
  Day 57: number analyzed (Participants) | 6 | 5 | 14
  Day 57 | 38 (30) | 27 (22) | 40 (31)
  Day 64: number analyzed (Participants) | 5 | 3 | 11
  Day 64 | 30 (29) | 30 (26) | 42 (35)
  Day 71: number analyzed (Participants) | 3 | 2 | 4
  Day 71 | 68 (33) | 63 (13) | 50 (34)
  Day 78: number analyzed (Participants) | 3 | 2 | 4
  Day 78 | 78 (39) | 105 (2) | 60 (26)
  Day 85: number analyzed (Participants) | 3 | 2 | 4
  Day 85 | 75 (38) | 64 (28) | 74 (24)
  Day 92: number analyzed (Participants) | 3 | 2 | 4
  Day 92 | 98 (42) | 95 (6) | 71 (23)
  Day 99: number analyzed (Participants) | 3 | 1 | 4
  Day 99 | 67 (11) | 89 (NA) — Only 1 participant contributed data at this time point. | 52 (16)
  Day 106: number analyzed (Participants) | 3 | 1 | 4
  Day 106 | 52 (34) | 43 (NA) — Only 1 participant contributed data at this time point. | 77 (28)
  Day 113: number analyzed (Participants) | 2 | 1 | 4
  Day 113 | 59 (15) | 53 (NA) — Only 1 participant contributed data at this time point. | 59 (7)
  Day 120: number analyzed (Participants) | 2 | 1 | 4
  Day 120 | 64 (34) | 59 (NA) — Only 1 participant contributed data at this time point. | 60 (16)

6. Secondary Outcome: Summary of Plasma Citrulline Levels Over Time
Description: Blood samples were collected at baseline, day 1 (pre-injection), day 4, day 8, and every 7 days thereafter for plasma citrulline levels.
Time Frame: Up to 9 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Number analyzed (Participants) | 6 | 5 | 19
uM
  Day 0: number analyzed (Participants) | 6 | 5 | 10
  Day 0 | 38 (17) | 29 (8) | 23 (14)
  Day 4 | 195 (89) | 158 (84) | 225 (106)
  Day 8 | 152 (40) | 121 (51) | 280 (125)
  Day 15: number analyzed (Participants) | 6 | 5 | 18
  Day 15 | 127 (71) | 125 (122) | 280 (150)
  Day 22: number analyzed (Participants) | 6 | 5 | 18
  Day 22 | 141 (102) | 174 (165) | 245 (175)
  Day 29: number analyzed (Participants) | 5 | 5 | 16
  Day 29 | 99 (59) | 126 (126) | 169 (148)
  Day 36: number analyzed (Participants) | 6 | 5 | 15
  Day 36 | 116 (75) | 104 (115) | 139 (149)
  Day 43: number analyzed (Participants) | 6 | 5 | 14
  Day 43 | 106 (81) | 135 (149) | 71 (72)
  Day 50: number analyzed (Participants) | 6 | 5 | 14
  Day 50 | 58 (31) | 77 (88) | 66 (76)
  Day 57: number analyzed (Participants) | 6 | 5 | 14
  Day 57 | 71 (51) | 47 (29) | 64 (76)
  Day 64: number analyzed (Participants) | 5 | 3 | 11
  Day 64 | 76 (80) | 108 (133) | 60 (54)
  Day 71: number analyzed (Participants) | 3 | 2 | 4
  Day 71 | 35 (9) | 19 (9) | 45 (34)
  Day 78: number analyzed (Participants) | 3 | 2 | 4
  Day 78 | 40 (12) | 44 (29) | 30 (19)
  Day 85: number analyzed (Participants) | 3 | 2 | 4
  Day 85 | 50 (30) | 23 (6) | 32 (11)
  Day 92: number analyzed (Participants) | 3 | 2 | 4
  Day 92 | 44 (21) | 27 (2) | 29 (18)
  Day 99: number analyzed (Participants) | 3 | 1 | 4
  Day 99 | 33 (13) | 31 (NA) — Only 1 participant contributed data at this time point. | 23 (12)
  Day 106: number analyzed (Participants) | 3 | 1 | 4
  Day 106 | 33 (21) | 33 (NA) — Only 1 participant contributed data at this time point. | 29 (10)
  Day 113: number analyzed (Participants) | 2 | 1 | 4
  Day 113 | 35 (12) | 22 (NA) — Only 1 participant contributed data at this time point. | 23 (10)
  Day 120: number analyzed (Participants) | 2 | 1 | 4
  Day 120 | 37 (14) | 47 (NA) — Only 1 participant contributed data at this time point. | 22 (8)

7. Secondary Outcome: Summary of ADI-PEG 20 Immunogenicity Over Time
Description: Blood samples were collected at baseline, day 1 (pre-injection), day 4, day 8, and every 7 days thereafter for detection of anti-ADI antibodies.
Time Frame: Up to 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log 10 U/mL
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Number analyzed (Participants) | 6 | 5 | 19
log 10 U/mL
  Day 0: number analyzed (Participants) | 6 | 5 | 10
  Day 0 | 0.2 (0.4) | 0.2 (0.5) | 0.1 (0.3)
  Day 4 | 0.2 (0.4) | 0.0 (0.0) | 0.4 (0.5)
  Day 8 | 0.2 (0.4) | 0.4 (0.5) | 0.4 (0.5)
  Day 15: number analyzed (Participants) | 6 | 5 | 18
  Day 15 | 0.5 (0.5) | 0.6 (0.5) | 0.8 (0.4)
  Day 22: number analyzed (Participants) | 6 | 5 | 18
  Day 22 | 0.5 (0.5) | 1.0 (0.6) | 0.7 (0.5)
  Day 29: number analyzed (Participants) | 5 | 5 | 16
  Day 29 | 0.8 (0.4) | 1.4 (0.5) | 1.3 (0.9)
  Day 36: number analyzed (Participants) | 6 | 5 | 15
  Day 36 | 0.8 (0.8) | 1.8 (0.4) | 1.9 (1.1)
  Day 43: number analyzed (Participants) | 6 | 5 | 14
  Day 43 | 1.2 (1.2) | 1.8 (0.4) | 2.4 (1.2)
  Day 50: number analyzed (Participants) | 6 | 5 | 14
  Day 50 | 1.5 (1.2) | 2.2 (0.4) | 2.9 (1.5)
  Day 57: number analyzed (Participants) | 6 | 5 | 14
  Day 57 | 1.5 (0.8) | 2.4 (0.5) | 3.0 (1.2)
  Day 64: number analyzed (Participants) | 5 | 3 | 11
  Day 64 | 2.0 (1.0) | 2.0 (0.0) | 3.0 (1.3)
  Day 71: number analyzed (Participants) | 3 | 2 | 4
  Day 71 | 2.3 (0.6) | 2.5 (0.7) | 3.5 (0.6)
  Day 78: number analyzed (Participants) | 3 | 2 | 4
  Day 78 | 2.7 (0.6) | 2.5 (0.7) | 4.0 (0.8)
  Day 85: number analyzed (Participants) | 3 | 2 | 4
  Day 85 | 2.7 (0.6) | 2.0 (0.0) | 4.0 (0.8)
  Day 92: number analyzed (Participants) | 3 | 2 | 4
  Day 92 | 3.0 (0.0) | 3.0 (0.0) | 4.0 (0.8)
  Day 99: number analyzed (Participants) | 3 | 1 | 4
  Day 99 | 3.0 (1.0) | 3.0 (NA) — Only 1 participant contributed data at this time point. | 3.8 (1.3)
  Day 106: number analyzed (Participants) | 3 | 1 | 4
  Day 106 | 3.0 (1.0) | 3.0 (NA) — Only 1 participant contributed data at this time point. | 4.0 (0.8)
  Day 113: number analyzed (Participants) | 2 | 1 | 4
  Day 113 | 3.0 (0.0) | 2.0 (NA) — Only 1 participant contributed data at this time point. | 4.0 (1.4)
  Day 120: number analyzed (Participants) | 2 | 1 | 4
  Day 120 | 3.0 (0.0) | 4.0 (NA) — Only 1 participant contributed data at this time point. | 4.5 (1.3)

8. Secondary Outcome: Correlation Between ASS Tumor Expression and Clinical Response
Description: Expression of ASS was analyzed by immunohistochemistry in tumor samples (archived or biopsy) at baseline and compared with overall best clinical response per RECIST. ASS tumor expression is categorized as either negative or ≤ 5% positive tumor cells.
Time Frame: Up to 12 months
Population: Includes all subjects who had an ASS antigen assay performed at Baseline
Measure: Number; unit: participants
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
Number analyzed (Participants) | 6 | 6 | 17
participants
  ≤5% Positive ASS & Progressive Disease | 2 | 0 | 3
  Negative ASS & Stable Disease | 1 | 1 | 0
  Negative ASS & Progressive Disease | 3 | 5 | 12
  Negative ASS & Missing Response | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs).
Description: AE documentation included onset/resolution dates, severity using NCI CTCAE (v4.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per subject at the maximum reported grade
Groups:
- Cohort 1: ADI-PEG 20 40 IU/m^2/Week: Includes subjects who received 40 IU/m^2/week of ADI-PEG 20
- Cohort 2: ADI-PEG 20 80 IU/m^2/Week: Includes subjects who received 80 IU/m^2/week of ADI-PEG 20
- Cohort 3: ADI-PEG 20 160 IU/m^2/Week: Includes subjects who received 160 IU/m^2/week of ADI-PEG 20
Arm/Group | Cohort 1: ADI-PEG 20 40 IU/m^2/Week | Cohort 2: ADI-PEG 20 80 IU/m^2/Week | Cohort 3: ADI-PEG 20 160 IU/m^2/Week
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 1/19
Serious Adverse Events (participants affected / at risk) | 4/6 | 1/6 | 6/19
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ADI-PEG 20 40 IU/m^2/Week (N=6) | Cohort 2: ADI-PEG 20 80 IU/m^2/Week (N=6) | Cohort 3: ADI-PEG 20 160 IU/m^2/Week (N=19)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphadenectomy (Surgical and medical procedures) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ADI-PEG 20 40 IU/m^2/Week (N=6) | Cohort 2: ADI-PEG 20 80 IU/m^2/Week (N=6) | Cohort 3: ADI-PEG 20 160 IU/m^2/Week (N=19)
Injection site pain (General disorders) | 2 | 1 | 11
Fatigue (General disorders) | 1 | 2 | 10
Nausea (Gastrointestinal disorders) | 4 | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 5
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Dizziness (Nervous system disorders) | 2 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Injection site rash (General disorders) | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Pyrexia (General disorders) | 1 | 0 | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Injection site erythema (General disorders) | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Injection site discomfort (General disorders) | 0 | 0 | 2
Injection site reaction (General disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Weight decreased (Investigations) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less